CLINICAL TRIAL: NCT03844243
Title: Interaction Between NGF and Exercise-induced Ischemia, and the Influence of the Pain Modulating System in a Prolonged NGF Sensitized Muscle.
Brief Title: Exercise-induced Ischemia and the Influence of Pain Modulation in a Nerve Growth Factor (NGF) Model
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Line Bay Sørensen, PhD.stud., Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N-2017-0007_S3
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pain Response; Hyperalgesia; Healthy Subjects
Keywords: NGF-induced hyperalgesia; Exercise-induced ischemic pain; Pain modulation; NGF pain model
MeSH Terms: conditions — Hyperalgesia | interventions — Nerve Growth Factor; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGF condition + Control condition (Experimental): All participants will receive 3 single injection of NGF (1ug/0.5ml) repeated over 3 separate days in their dominant tibialis anterior muscle.
  After 4 weeks:
  All participants will receive 3 single injection of isotonic-saline (9%/0.5ml) repeated over 3 separate days in their dominant tibialis anterior muscle.
  Interventions: Drug: NGF; Drug: Isotonic-saline
- Control condition + NGF condition (Experimental): All participants will receive 3 single injection of isotonic-saline (9%/0.5ml) repeated over 3 separate days in their dominant tibialis anterior muscle.
  After 4 weeks:
  All participants will receive 3 single injection of NGF (1ug/0.5ml) repeated over 3 separate days in their dominant tibialis anterior muscle.
  Interventions: Drug: NGF; Drug: Isotonic-saline

INTERVENTIONS:
Drug: NGF — Intramuscular injection
  Other Names: Beta-Nerve Growth Factor, Human
Drug: Isotonic-saline — Intramuscular injection
  Other Names: Control

SUMMARY:
The purpose of this study is to investigate responses of pain and the maintenance of mechanical muscle hypersensitivity following an acute exercise-induced ischemic condition repeated over time in a prolonged NGF-sensitized muscle. Additionally, the influence of the pain modulating system on prolonged NGF muscle hypersensitivity caused by peripheral mechanisms and central mechanisms will also be investigated.

DETAILED DESCRIPTION:
The hypothesis is that an ischemic conditioning in a NGF-sensitized muscle is able to facilitate pain responses and that over time the pain modulation system is responsible for a subsequent reduction in muscle sensitivity towards mechanical pressure and a decrease in pain intensity following a period of NGF-induced muscle hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and pain free volunteers

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, mental illnesses, or psychiatric diseases.
* Past history of chronic pain in the musculoskeletal system (muscle, joint, cartilage, connective tissue)
* Participation in other pain trials throughout the study period
* Lack of ability to cooperate
* Taking any analgesic 24 hours before the injections
* Performing any strenuous leg exercise through out the study period causing sore muscles

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-18 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle pain sensitivity (PPTs values) assessed by pressure algometer | Change from baseline at 3 week
  Pressure pain thresholds (PPTs) are assessed over the dominant tibialis anterior muscle using a handhold pressure algometer.

SECONDARY OUTCOMES:
Ischemic-induced pain intensity | Assessed right after the exercise has been performed, change from baseline at 3 weeks
  Subjects perform a repeated static exercise with their dominant leg while a cuff is mounted over the knee to occlude the blodflow from the muscle (ischemia). Subjects subsequently rate their perceived pain intensity verbally on a 11-point numeric rating scale (NRS) rating from 0 (no pain) to 10 (worst pain imaginable).
Functional muscle pain | Change from baseline at 3 weeks
  Subjects evaluate their muscle pain during movement using a 7-point Likert Scale for lower limp rating from 0 (a complete absence of pain) to 6 (a severe pain that limits my ability to move).
Conditioning pain modulation (CPM) efficacy | Change from baseline at 3 weeks
  A test stimuli will be applied and compared with a test stimuli simultaneous a condition stimuli.
Temporal summation of pain | Change from baseline at 3 weeks
  10 repeated stimuli will be applied and subjects will be asked to rate the pain for each individual stimuli on a 11-point visual analogue scale (VAS) rating from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Line Bay Sørensen, PhD. stud., Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No